CLINICAL TRIAL: NCT01140971
Title: TRANSCERVICAL FOLEY CATHETER (FOLEY) Versus INTRAVAGINAL MISOPROSTOL FOR CERVICAL RIPENING AND INDUCTION OF LABOR: A RANDOMIZED CLINICAL TRIAL.
Brief Title: Foley Catheter Versus Vaginal Misoprostol for Cervical Ripening and Induction of Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Municipal Hospital Vila Nova Cachoeirinha (Other)
Responsible Party: Nelson Sass, Maternidade Escola de Vila Nova Cachoeirinha
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MHVNCachoeirinha
Record Dates: First submitted 2010-06-08; First posted 2010-06-10 (Estimated); Last update posted 2010-06-10 (Estimated); Status verified 2009-09

CONDITIONS: Pregnancy, Prolonged; Pre Eclampsia; Oligohydramnios
Keywords: Balloon dilatation,; misoprostol,; cervical ripening,; obstetric labor,; labor induced.
MeSH Terms: conditions — Pregnancy, Prolonged; Pre-Eclampsia; Oligohydramnios | interventions — Misoprostol; Urinary Catheterization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Misoprostol (Active Comparator): Use 25 micrograms vaginal every 6 hours (max dosis 200 micrograms in 48 hours)
  Interventions: Drug: Misoprostol
- Foley (Active Comparator): Foley catheter number 14 or 16 was installed intracervical for no more than 48 hours.
  Interventions: Device: Foley

INTERVENTIONS:
Drug: Misoprostol — Vaginal application of 25 micrograms every 6 hours until cervical ripening reach Bishop 6 or more
  Other Names: Prostokos 25 micrograms
  Arms: Misoprostol
Device: Foley — After Foley introduction, every 6 hours vaginal exam was performed. The cases on Bishop score increase or occurred spontaneous exit of catheter or spontaneous labour had been initiated are considered success.The failure was adopted if after48 hours occurred no cervical modifications.
  Arms: Foley

SUMMARY:
PURPOSE: The purpose of this study is to determine the effectiveness of balloon dilatation (Foley) with vaginal misoprostol for cervical ripening and induction of labor.

METHOD: a randomized clinical assay has been performed with 160 women with indication of induction of labor, randomly divided in two groups, 80 for Foley catheter and 80 for misoprostol.

DETAILED DESCRIPTION:
The cesarean delivery rate has risen dramatically in almost all world. Brazil shows the highest rate in the world so we need urgently efforts to reduce this fact. Several studies have shown that maternal morbidity and mortality rates are higher in cesarean deliveries. On the other hand an abdominal delivery cost much more than a vaginal delivery.

A clinical trial to assess the performance of two simple and sheep methods can provide evidence based on local experience. Our results alow us to recommend both methods for clinical practice with a good possibility to reduce cesarean rates and without adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age from 37 weeks,
* feto unic, alive and cephalic,
* Bishop index equal or lesser than four.

Exclusion Criteria:

* uterine scar,
* premature rupture of the membranes,
* fetal weight bigger than 4000 g,
* previous placenta,
* conditions that imposed the immediate ending of the gestation.

Ages: 19 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2006-01; Primary Completion 2008-03 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Cervical ripening | 48 hous after start the method
  Foley Group: catheter stay no more that 48 hours. Every 6 hours vaginal exam was performed. The cases on Bishop score increase or occurred spontaneous exit of catheter or spontaneous labour had been initiated are considered success.The failure was adopted if after48 hours occurred no cervical modifications.
  Misoprostol group: was introduced 25 microgram every 6 hour (max 200microg)if cervical conditions were unchanged. In the case of cervical evolution or start of labour the method was considered success.The failure was adopted if after 48 there was no cervical modifications.

SECONDARY OUTCOMES:
Cesarean | The action of methods were assessed for 48 hours after start.
  After 48 hours if there was no cervical ripening or espontaneous labor the case was classified as failure of method and a cesarean was performed
Need of oxytocin | 48 hours after start method
  In cases on the cervical ripening had occurred but the spontaneous labor not start.
need of neonatal intensive care | 7 first days after birth
  The condition of babies at birth and needs of intensive care as mechanic ventilation or others interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Nelson Sass, pHD, Principal Investigator — Maternidade Escola de Vila Nova Cachoeirinha
Locations (1):
- MHVNCachoeirinha, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Sciscione AC, Muench M, Pollock M, Jenkins TM, Tildon-Burton J, Colmorgen GH. Transcervical Foley catheter for preinduction cervical ripening in an outpatient versus inpatient setting. Obstet Gynecol. 2001 Nov;98(5 Pt 1):751-6. doi: 10.1016/s0029-7844(01)01579-4. PMID 11704164
- [Background] Afolabi BB, Oyeneyin OL, Ogedengbe OK. Intravaginal misoprostol versus Foley catheter for cervical ripening and induction of labor. Int J Gynaecol Obstet. 2005 Jun;89(3):263-7. doi: 10.1016/j.ijgo.2005.02.010. Epub 2005 Apr 2. PMID 15919393
- [Background] Boulvain M, Kelly A, Lohse C, Stan C, Irion O. Mechanical methods for induction of labour. Cochrane Database Syst Rev. 2001;(4):CD001233. doi: 10.1002/14651858.CD001233. PMID 11687101